CLINICAL TRIAL: NCT05005936
Title: Comparing the Performance of Automated Breast Ultrasonography (ABUS) to Hand-Held Breast Ultrasonography (WBUS) in Breast Cancer Treatment Response Assessment in a Tertiary Cancer Center: A Prospective Study
Brief Title: Comparing the Performance of Automated Breast Ultrasonography to Hand-Held Whole Breast Ultrasonography in Breast Cancer Treatment Response Assessment
Status: Withdrawn | Type: Observational
Why Stopped: No participants Enrolled
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0831; NCI-2021-05381 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0831 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-30; First posted 2021-08-16 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (ABUS, WBUS): Patients undergo ABUS over 15 minutes followed by WBUS over 30 minutes at baseline, mid-treatment and pre-surgery (end of treatment).
  Interventions: Procedure: Ultrasonography

INTERVENTIONS:
Procedure: Ultrasonography — Undergo ABUS
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasound; Ultrasound Imaging; Ultrasound Test; Ultrasound, Medical; US
Procedure: Ultrasonography — Undergo WBUS
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasound; Ultrasound Imaging; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This study compares the performance of automated breast ultrasonography and conventional hand-held whole breast ultrasonography when checking for response to breast cancer treatment. Breast ultrasonography is operator dependent and time-intensive. Automated breast ultrasonography scanners were developed to allow standardization of ultrasound scanning and scanning to be performed by any technologist, with or without previous ultrasound experience, without physician involvement. This study may validate the use of the automated breast ultrasonography.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate and compare the accuracy of automated breast ultrasonography (ABUS) and hand-held whole breast ultrasonography (WBUS) in predicting pathology complete response (pCR) with relative tumor volume change, using the receiver operating characteristic (ROC) curve analysis.

SECONDARY OBJECTIVES:

I. To evaluate the reproducibility of tumor volume measurements obtained by ABUS and handheld WBUS, respectively, using data collected at baseline for initial staging.

II. To assess the agreement in relative tumor volume change (RC) (end-of-treatment versus [vs.] pre-treatment) between ABUS and WBUS.

III. To estimate and compare the following diagnostic measures for ABUS and WBUS: sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

OUTLINE:

Patients undergo ABUS over 15 minutes followed by WBUS over 30 minutes at baseline, mid-treatment and pre-surgery (end of treatment).

ELIGIBILITY:
Inclusion Criteria:

* The subjects to be studied will include patients seen in MD Anderson Breast imaging clinic at the Texas Medical Center (TMC)
* With breast cancer or suspicion of breast cancer
* Male or female who is older than 18 years of age
* Of any race
* Who consent to obtain technologist performed breast ultrasound and automated breast ultrasound
* English and non-English speakers (with language interpreter to assist in translation for non-English speakers)

Exclusion Criteria:

* Patient who is less than 18 years of age
* Imaging obtained outside of MD Anderson TMC
* Surgery pathology from outside of MD Anderson will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer or suspicion of breast cancer seen in MD Anderson Breast imaging clinic at the Texas Medical Center (TMC)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic (ROC) curve | through study completion, an average of 1 year
  Will compute relative tumor volume change for both automated breast ultrasonography (ABUS) and hand-held whole breast ultrasonography (WBUS) and estimate pathology complete response ROC curves for each. Will estimate the areas under the ROC curves along with 95% confidence intervals and then compare the values statistically.

SECONDARY OUTCOMES:
Tumor volume | through study completion, an average of 1 year
  Will compute the intraclass correlation coefficient for each method along with 95% confidence intervals and then compare these estimates.
Relative tumor volume change | through study completion, an average of 1 year
  Will compute the relative change in tumor volume for ABUS and WBUS and assess their agreement using the Bland-Altman approach.
Sensitivity | through study completion, an average of 1 year
  The cutoff point will be determined using Youden Index, i.e., the point that maximize (sensitivity specificity).
Specificity | through study completion, an average of 1 year
  The cutoff point will be determined using Youden Index, i.e., the point that maximize (sensitivity specificity).
Positive predictive value | through study completion, an average of 1 year
Negative predictive value | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Monica L Huang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://mdanderson.org